CLINICAL TRIAL: NCT00267475
Title: Clinical and Immunological Evaluation of Eosinophil Associated Gastrointestinal Disorders (EGID)
Brief Title: Data Bank for Eosinophilic Disorders
Status: Completed | Type: Observational
Sponsor: Marc Rothenberg (Other)
Responsible Party: Sponsor-Investigator, Marc Rothenberg, MD, PhD, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Other Study IDs: 01-3-15; CSA1002171
Record Dates: First submitted 2005-12-15; First posted 2005-12-21 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-01

CONDITIONS: Eosinophilic Esophagitis; Gastritis; Enteritis; Eosinophilic Colitis; Eosinophilic Gastroenteritis
Keywords: eosinophilic esophagitis; eosinophilic gastritis; eosinophilic enteritis; eosinophilic colitis; eosinophilic gastroenteritis
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastritis; Enteritis; Eosinophilic enteropathy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to conduct a translational study in patients with primary eosinophil associated gastrointestinal disorders [EGID] (e.g. eosinophilic esophagitis eosinophilic gastritis, eosinophilic enteritis [EE], eosinophilic colitis, and eosinophilic gastroenteritis [EGE]) with the aim of developing a data bank containing pertinent patient demographic information, tissue samples, and DNA, which will facilitate research on the pathophysiology of inflammatory disorders and the development of a verified successful clinical treatment program.

ELIGIBILITY:
Patients with an eosinophil associated gastrointestinal disorder (EGID), family members of patients with EGID, or normal controls.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with an eosinophilic disorder and patients without an eosinophilic disorder to serve as normal controls
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2001-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E. Rothenberg, M.D., Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States